CLINICAL TRIAL: NCT02375204
Title: A Randomized Phase III Trial Comparing Conventional-Dose Chemotherapy Using Paclitaxel, Ifosfamide, and Cisplatin (TIP) with High-Dose Chemotherapy Using Mobilizing Paclitaxel Plus Ifosfamide Followed by High-Dose Carboplatin and Etoposide (TI-CE) As First Salvage Treatment in Relapsed or Refractory Germ Cell Tumors
Brief Title: Standard-Dose Combination Chemotherapy or High-Dose Combination Chemotherapy and Stem Cell Transplant in Treating Patients with Relapsed or Refractory Germ Cell Tumors
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); European Organisation for Research and Treatment of Cancer - EORTC (Network); Movember Foundation (Other); Institute of Cancer Research (ICR), United Kingdom (Unknown); Cancer Research UK (Other); UNICANCER (Other); Irish Group CTI (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A031102; U10CA180821 (NIH); NCI-2014-01696 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2015-02-20; First posted 2015-03-02 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Germ Cell Tumor; Teratoma; Choriocarcinoma; Germinoma; Mixed Germ Cell Tumor; Yolk Sac Tumor; Childhood Teratoma; Malignant Germ Cell Neoplasm; Extragonadal Seminoma; Non-seminomatous Germ Cell Tumor; Seminoma
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Teratoma; Choriocarcinoma; Germinoma; Endodermal Sinus Tumor; Nonseminomatous germ cell tumor; Seminoma | interventions — Paclitaxel; Ifosfamide; Cisplatin; Granulocyte Colony-Stimulating Factor; Carboplatin; etoposide phosphate; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: TIP (Other): Patients will receive treatment for 4 cycles administered every 21 days.
  Cycles 1-4 (1 cycle = 21 days)
  * paclitaxel 250 mg/m^2 IV over 24 hours on Day 1 including premedication as defined in the protocol (eg, dexamethasone, diphenhydramine and H2 blocker)
  * ifosfamide 1500 mg/m^2 IV daily on Days 2-5 with mesna protection as defined in the protocol
  * cisplatin 25 mg/m^2 IV daily on Days 2-5
  * pegylated G-CSF 6 mg subcutaneous on Day 6 or 7 or G-CSF as defined in the protocol on Days 6-18
  Patients may commence with each Arm A cycle provided they meet the criteria as defined in the protocol.
  Interventions: Drug: paclitaxel; Drug: ifosfamide; Drug: cisplatin; Drug: pegylated G-CSF; Drug: G-CSF
- Arm B: TI-CE (Other): Patients will receive treatment for a total of 5 cycles.
  Cycles 1-2 (1 cycle = 14 days)
  * paclitaxel 200 mg/m^2 IV over 3 hours on Day 1 including premedication as defined in the protocol (eg, dexamethasone, diphenhydramine and H2 blocker)
  * ifosfamide 2000 mg/m^2 IV daily on Days 1-3 with mesna protection as defined in the protocol
  * G-CSF 10 µg/kg subcutaneously on Days 3-15 (cycle 1) and Days 3-14 (cycle 2) or pegylated G-CSF 6 mg subcutaneous on Day 4 or 6 (cycle 1) and Day 4 or 5 (cycle 2)
  * leukapheresis every 14 days, if there is an inadequate number of CD34+ cells/kg collected in cycle 1
  Cycles 3-5 (1 cycle = 21 days)
  * carboplatin daily on Days 1-3
  * etoposide 400 mg/m^2 daily on Days 1-3
  * stem cell reinfusion on day 5
  * pegylated G-CSF 6 mg subcutaneously or G-CSF at approximately 5 µg/kg daily on Days 5-15
  Patients may commence with each Arm B cycle provided they meet the criteria as defined in the protocol.
  Interventions: Drug: paclitaxel; Drug: ifosfamide; Drug: pegylated G-CSF; Drug: G-CSF; Drug: carboplatin; Drug: etoposide phosphate; Procedure: stem cell reinfusion

INTERVENTIONS:
Drug: paclitaxel — IV
  Other Names: Taxol
Drug: ifosfamide — IV
  Other Names: Ifex®, IFOS
Drug: cisplatin — IV
  Other Names: CDDP
  Arms: Arm A: TIP
Drug: pegylated G-CSF — IV
Drug: G-CSF — IV
Drug: carboplatin — IV
  Other Names: Paraplatin®, CBDCA
  Arms: Arm B: TI-CE
Drug: etoposide phosphate — IV
  Other Names: VePesid®, Toposar®, VP16
  Arms: Arm B: TI-CE
Procedure: stem cell reinfusion — surgical procedure
  Arms: Arm B: TI-CE

SUMMARY:
This randomized phase III trial studies how well standard-dose combination chemotherapy works compared to high-dose combination chemotherapy and stem cell transplant in treating patients with germ cell tumors that have returned after a period of improvement or did not respond to treatment. Drugs used in chemotherapy, such as paclitaxel, ifosfamide, cisplatin, carboplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as filgrastim or pegfilgrastim, and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. It is not yet known whether high-dose combination chemotherapy and stem cell transplant are more effective than standard-dose combination chemotherapy in treating patients with refractory or relapsed germ cell tumors.

DETAILED DESCRIPTION:
The study is an international collaboration with European sites. Collaborators on the study include the National Cancer Institute, the European Organization for Research and Treatment of Cancer and the Movember Foundation. Randomization will be stratified by region (North America and Europe) and by modified IPFSG (International Prognostic Factor Study Group) risk classification (low, intermediate and high). The primary and secondary objectives are described below.

Primary Objective:

1. To compare the overall survival in patients treated with conventional-dose chemotherapy using the TIP regimen with high-dose chemotherapy (HDCT) plus autologous stem cell transplant (ASCT) using the TI-CE regimen as initial salvage treatment of patients with relapsed or refractory germ cell tumors (GCT)

Secondary Objectives:

1. To compare the progression-free survival (PFS) of patients treated with initial salvage HDCT with TI-CE versus initial salvage CDCT with TIP
2. To compare the favorable response rate (FRR) of patients treated with initial salvage HDCT with TI-CE versus initial salvage CDCT with TIP
3. To compare the toxicity, including treatment-related mortality, associated with high-dose chemotherapy and ASCT using TI-CE compared with conventional-dose chemotherapy using TIP as initial salvage treatment for patients with relapsed or refractory GCT
4. To prospectively evaluate the IPFSG scoring system as a predictor of outcome to initial salvage therapy in patients with relapsed or refractory GCT. In this trial, randomization will be stratified by a modification of their IPFSG category and we will prospectively evaluate whether or not actual outcomes vary by risk group in the appropriate manner (low risk patients have higher OS than high-risk group).
5. To evaluate the association between tumor marker decline rates of Alpha-Fetoprotein (AFP) and Human Chorionic Gonadotropin (HCG) with OS and PFS.

Treatment is to continue until disease progression, unacceptable toxicity or completion of all protocol treatment.

ELIGIBILITY:
1. Documentation of Disease

   * Histologic Documentation: Confirmation of GCT histology (both seminoma and nonseminoma) on pathologic review at the center of enrollment.
   * Tumor may have originated in any primary site. NOTE: In rare circumstances, patients will be allowed to enroll even if a pathologic diagnosis may not have been established.
   * This would require a clinical situation consistent with the diagnosis of GCT (testicular, peritoneal, retroperitoneal or mediastinal mass, elevated tumor marker levels {HCG ≥ 500; AFP ≥ 500} and typical pattern of metastases)
2. Evidence of Disease

   * Must have evidence of progressive or recurrent GCT (measurable or non-measurable) following one line of cisplatin-based chemotherapy, defined as meeting at least one of the following criteria:

     * Tumor biopsy of new or growing or unresectable lesions demonstrating viable non-teratomatous GCT (enrollment on this study for adjuvant treatment after macroscopically complete resection of viable GCT is not allowed). In the event of an incomplete gross resection where viable GCT is found, patients will be considered eligible for the study.
     * Consecutive elevated serum tumor markers (HCG or AFP) that are increasing. Increase of an elevated LDH alone does not constitute progressive disease.
     * Development of new or enlarging lesions in the setting of persistently elevated HCG or AFP, even if the HCG and AFP are not continuing to increase.
3. Prior Treatment

   * Must have received 3-6 cycles of cisplatin-based chemotherapy as part of first-line (initial) chemotherapy.

     * Prior POMBACE, CBOP-BEP, or GAMEC are allowed.
     * Note: For patients requiring immediate treatment, 1 cycle of conventional-dose salvage chemotherapy is allowed. Therefore, these patients may have received 7 prior cycles of chemotherapy. 6 cycles as part of first-line chemotherapy and 1 cycle of salvage conventional chemotherapy.
   * No more than one prior line of chemotherapy for GCT (other than the 1 cycle of salvage chemotherapy as defined in the protocol)

     * Definition of one line of chemotherapy: One line of therapy can in some cases consist of 2 different cisplatin-based treatment combinations, provided there is no disease progression between these two regimens.
     * Prior treatment with carboplatin as adjuvant therapy is allowed, provided patients meet other eligibility criteria (e.g., the patient has also received 3-4 cycles of cisplatin-based chemotherapy).
     * Prior treatment with 1-2 cycles of BEP or EP as adjuvant chemotherapy for early stage GCT is allowed, provided the patient also received 3-4 cycles of BEP or EP again at relapse. Patients treated with 3-4 cycles of VIP at relapse following 1-2 cycles of BEP/EP are not eligible as this would be considered more than 1 line of prior therapy.
   * No prior treatment with high-dose chemotherapy (defined as treatment utilizing stem cell rescue)
   * No prior treatment with TIP with the exception when given as a bridge to treatment on protocol for patients with rapidly progressive disease who cannot wait to complete the eligibility screening process. Only one cycle is allowed.
   * No concurrent treatment with other cytotoxic drugs or targeted therapies.
   * No radiation therapy (other than to the brain) within 14 days of day 1 of protocol chemotherapy except radiation to brain metastases, which must be completed 7 days prior to start of chemotherapy.
   * No previous chemotherapy within 17 days prior to enrollment. A minimum of three weeks after the last day of the start of the previous chemotherapy regimen before the first day of chemotherapy on study protocol.
   * Must have adequate recovery from prior surgery (eg, healed scar, resumption of diet)
4. Age ≥ 14 years (≥ 18 years in Germany)
5. ECOG Performance Status 0 to 2
6. Male gender
7. Required Initial Laboratory Values:

   * Absolute Neutrophil Count (ANC) ≥ 1,500/mm^3
   * Platelet Count ≥ 100,000/mm^3
   * Calculated creatinine clearance ≥ 50 mL/min
   * Bilirubin ≤ 2.0 x upper limits of normal (ULN)
   * AST/ALT ≤ 2.5 x upper limits of normal (ULN)
8. No concurrent malignancy other than non-melanoma skin cancer, superficial noninvasive (pTa or pTis) TCC of the bladder, contralateral GCT, or intratubular germ cell neoplasia. Patients with a prior malignancy, but at least 2 years since any evidence of disease are allowed.
9. Negative Serology (antibody test) for the following infectious diseases:

   * Human Immunodeficiency Virus (HIV) type 1 and 2
   * Human T-cell Leukemia Virus (HTLV) type 1 and 2 (mandatory in US but optional in Canada and Europe)
   * Hepatitis B surface antigen
   * Hepatitis C antibody
10. No late relapse with completely surgically resectable disease. Patients with late relapses (defined as relapse ≥ 2 years from the date of completion of the last chemotherapy regimen) whose disease is completely surgically resectable are not eligible. Patients with late relapses who have unresectable disease are eligible.
11. No large (≥ 2 cm) hemorrhagic or symptomatic brain metastases until local treatment has been administered (radiation therapy or surgery). Treatment may begin ≥ 7 days after completion of local treatment. Patients with small (< 2 cm) and asymptomatic brain metastases are allowed and may be treated with radiation therapy and/or surgery concurrently with Arm A or cycles 1 and 2 of Arm B if deemed medically indicated.

    Radiation therapy should not be given concurrently with high-dose carboplatin or etoposide.
12. No secondary somatic malignancy arising from teratoma (e.g., teratoma with malignant transformation) when it is actively part of the disease recurrence or progression.

Min Age: 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | Up to 36 months post-treatment

SECONDARY OUTCOMES:
progression free survival | Up to 36 months post-treatment
proportion of patients achieving either a complete response (CR) or partial response | Up to 3 months post-registration
treatment related mortality | Up to 30 days post-treatment
number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 3 months post-registration
Validation of International Prognostic Factor Study Group stratification system (eg, primary site, prior response, progression free interval) | Up to 3 years post-registration

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (125):
- United States (77):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - El Paso Children's Hospital, El Paso, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - University Hospital Saint Luc, Brussels
- Rigshospitalet University Hospital, Copenhagen, Denmark
- France (7):
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Tenon/Assistance Publique - Hopitaux de Paris, Paris
  - CHRU Strasbourg - Hospital Civil, Strasbourg
  - Center Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (11):
  - Technical University Dresden, Dresden, Saxony
  - University of Berlin Charite Campus Benjamin Franklin, Berlin
  - University of Dusseldorf, Düsseldorf
  - University of Essen, Essen
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - UniversitaetsKlinikum Heidelberg, Heidelberg
  - GK-Mittelrhein Saint Martin's, Koblenz
  - Philipps University Marburg, Marburg
  - Rotkreuzklinikum Munchen, Munich
  - Klinikum Nurnberg Nord, Nuremberg
  - University Hospital Ulm, Ulm
- Saint James Hospital, Dublin, Ireland
- Italy (4):
  - Ospedale di Circolo di Busto Arsizio, Busto Arsizio
  - Istituto Scientifico Romagnolo, Meldola
  - Istituto Nazionale Tumori, Milan
  - San Matteo Hospital, Pavia
- Netherlands (3):
  - The Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud University Nijmegen Medical Centre, Nijmegen
- Spain (4):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Duran i Reynals Hospital-Catalan Institute of Oncology, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
- Switzerland (3):
  - Inselspital, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - University Hospital Zurich, Zurich
- United Kingdom (8):
  - Saint Bartholomew's Hospital, London, England
  - Christie Hospital, Manchester, England
  - Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Saint James's University Hospital, West Yorkshire, England
  - Beatson Oncology Center, Glasgow, Scotland
  - Nottingham City Hospital, Nottingham
  - The Royal Marsden NHS Foundation Trust - Sutton, Surrey

REFERENCES:
- [Derived] Gleeson JP, Knezevic A, Bromberg M, Patil S, Sheinfeld J, Carver BS, Bains M, Jones DR, Bajorin DF, Bosl GJ, McHugh DJ, Funt SA, Motzer RJ, Feldman DR. Paclitaxel, Ifosfamide, and Cisplatin as Initial Salvage Chemotherapy for Germ Cell Tumors: Long-Term Follow-Up and Outcomes for Favorable- and Unfavorable-Risk Disease. J Clin Oncol. 2024 Sep 10;42(26):3130-3139. doi: 10.1200/JCO.23.02542. Epub 2024 Jul 19. PMID 39028926
- [Derived] Tan YY, Al-Bubseeree B, Irvine D, MacDonald G, McQuaker G, Parker A, Waterston A, White J. High-Dose Chemotherapy in Relapsed or Refractory Metastatic Germ-Cell Cancer: The Scotland Experience. Clin Genitourin Cancer. 2019 Apr;17(2):125-131. doi: 10.1016/j.clgc.2018.11.013. Epub 2018 Nov 17. PMID 30563754